CLINICAL TRIAL: NCT01129076
Title: Perceptions of Thalassemia Major in Singapore: An Exploratory Study of Stigma
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910104; 10-HG-N104
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-01-07

CONDITIONS: Thalassemia Major
Keywords: Thalassemia Major; Stigma; Singapore; Qualitative
MeSH Terms: conditions — beta-Thalassemia; Social Stigma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Thalassemia major (TM) is a chronic disorder that affects a person s ability to produce hemoglobin, resulting in anemia. Hemoglobin is a component of red blood cells that carries oxygen and nutrients to cells in the body. As a result, individuals require life-long blood transfusions and extensive medical management. Studies have shown that because of its demanding nature, TM might negatively affect an individual s quality of life, sense of self, and social integration, but little is known about affected individuals overall experiences with and perceptions of TM.
* TM is caused by a genetic change in the thalassemia gene. The disease is passed to children by parents who carry one copy of the altered thalassemia gene. The parents are called carriers of the condition and have a 25 percent chance of having a child with TM. It is possible to screen for carriers of TM and use this information for pregnancy planning and management.
* TM is common among people from South and South East Asia and is an important public health concern in Singapore. More research is needed to explore the lives of people with TM, and the societal perceptions that exist in Singapore about TM.

Objectives:

* To describe the familial, social, and professional experiences of individuals with TM.
* To investigate the social messages being given out about TM in Singapore and the sources of those messages.
* To explore the impact of these experiences, perceptions, and social messages on individuals who have TM.
* To explore how the experiences and perceptions of individuals who have TM affect their life, sense of self, social integration, and compliance with medical treatment.

Eligibility:

* Residents of Singapore who are 14 years of age or older, can speak English, and currently have TM.
* Parents of individuals with TM who are 14 years of age or older. Parents must be 21 years of age or older, be able to speak English, and have had caregiving responsibilities for their child at some point.

Design:

* All participants will have a one-time semi-structured interview, followed by a questionnaire to obtain demographic information.
* Interviews will be conducted in Singapore and are expected to last for 30 to 90 minutes.
* Individuals with TM will be asked about their own perceptions of TM; familial, social, and professional experiences involving TM; and their perceptions of others views and of social messages related to TM.
* Parents of individuals with TM will be asked about their experiences in caring for a child with TM, talking to their child about TM, telling people about their child s TM, and interacting with health care providers.

DETAILED DESCRIPTION:
Thalassemia major (TM) is a chronic, inherited hematological disorder that can require life-long medical care. As a result of the chronic and demanding nature of the condition, studies have shown that TM might negatively affect an individual s quality of life, sense of self, social integration, and compliance with medical treatment. Yet, little is known about affected individuals overall experiences with and perceptions of TM. In this study, the concept of stigma will be used to explore and understand these experiences and perceptions in the population of individuals with TM in Singapore. This study will involve qualitative interviews with TM patients and parents of TM patients. Interviews will focus on individuals family, social and professional experiences with TM; the social messages that exist in Singapore about TM and their sources; individuals perceptions of how others view TM; individuals own perceptions of TM; and the impact of these various experiences, messages and perceptions on the individual with TM. Interviews will be conducted with approximately 20-30 individuals with TM, and 10-20 parents of individuals with TM. Interviews will be transcribed and subjected to thematic analysis to identify common themes. The results of this study will further our understanding of the psychosocial burden of TM and the potential role of stigma in this population, which may ultimately inform the care for individuals with TM. The study s setting will also provide insights into the impact of the Singaporean sociocultural context on the psychosocial elements of living with a genetic condition, which might eventually help to inform the development of appropriate psychosocial support services and genetic counseling services in the region.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals who currently have TM and receive at least 8 blood transfusions in a year
* Residents of Singapore
* Must speak English
* Parents of individuals with TM will be eligible for participation if they are age 21 years or older
* Parents must be residents of Singapore
* Parents must speak English
* For a parent to participate in the study, it will not be required that his or her child also participate in the study or vice versa.

EXCLUSION CRITERIA:

* Children under age 14 years
* Non-English speaking individuals

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04-23; Study Completion 2016-01-07

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- Singapore (2):
  - Singapore General Hospital Outram Rd., Singapore
  - KK Women's & Children's Hospital, Singapore

REFERENCES:
- [Background] Ismail A, Campbell MJ, Ibrahim HM, Jones GL. Health Related Quality of Life in Malaysian children with thalassaemia. Health Qual Life Outcomes. 2006 Jul 2;4:39. doi: 10.1186/1477-7525-4-39. PMID 16813662
- [Background] Hoedemaekers R, ten Have H. Geneticization: the Cyprus paradigm. J Med Philos. 1998 Jun;23(3):274-87. doi: 10.1076/jmep.23.3.274.2585. PMID 9736189
- [Background] Major B, O'Brien LT. The social psychology of stigma. Annu Rev Psychol. 2005;56:393-421. doi: 10.1146/annurev.psych.56.091103.070137. PMID 15709941